Original Title of Study: L-methylfolate supplementation to OROS-methylphenidate pharmacotherapy in ADHD Adults: A double-blind, placebo-controlled, randomized clinical trial.

NCT Number: NCT01853280

Date of SAP Plan: 12/22/2016

## <u>Deplin Statistical Analysis Plan – Paper 1</u>

# 1. General Analysis Details

a. Analyses will be intention to treat and include all subjects that received deplin or placebo for at least 1 week. We will perform a per protocol analysis as a secondary analysis.

## 2. Demographic Characteristics & Baseline Efficacy Measures

- a. We will compare demographic characteristics and baseline efficacy measures between those randomized to placebo and those randomized to deplin to ensure that the randomization process was successful.
  - i. We will compare the groups using standard parametric and non-parametric tests (Student's t-test, Wilcoxon rank sum test, Pearson's chi-square test, Fisher's exact test).
  - i. Demographic characteristics will include age, gender, race, and socioeconomic status.
  - ii. Baseline efficacy measures will include AISRS, CGI, BRIEF-A GEC subscale, and GAF.

## 3. Safety

- a. Individual Adverse Events
  - i. We will report a frequency table of recurrent adverse events. No statistical analyses will be performed on individual AEs.
- b. Total Number of Adverse Events
  - i. We will compare the total number of AEs in each group using a Poisson regression model, which is the appropriate model for count data.
- c. Time-course of Adverse Events
  - i. We will analyze the time-course of AEs using a mixed effects Poisson model that predicts the total number of AEs from the drug group, study week, and drug group x study week interaction. The interaction will tell us if there is a difference in the occurrence of AEs between the groups over the course of the study.

#### d. Vitals

i. We will analyze vital signs using mixed effects regression models with the drug group, study week, and drug group x study week interaction as predictors.

#### 4. Primary Efficacy Measure (AISRS)

- a. We will analyze the AISRS using a mixed effects Poisson model that includes the drug group, study week, and drug group x study week interaction as predictors. Using this model is consistent with how we have analyzed the AISRS in previous publications.
  - i. If there are statistically significant differences in demographic characteristics or baseline efficacy measures then we will add variables to the model to control for them.

#### 5. Secondary Efficacy Measures

- a. Secondary outcomes measures will include the following: CGI, BRIEF-A, GAF, DESR, HAM-A, HAM-D, ASR, and CANTAB
  - i. We will analyze the GAF and BRIEF-A using mixed effects Poisson models that include the drug group, study week, and drug group x study week interaction as predictors.
  - ii. We will analyze the CGI using a mixed effects ordinal logistic regression model that includes the drug group, study week, and drug group x study week interaction as predictors.
  - iii. For the DESR, HAM-A, HAM-D, ASR, CANTAB, and BRIEF-A, subjects will be define as having normal or abnormal scores based on pre-defined cutoffs from the literature. We will analyze these outcomes using mixed effects logistic regression models that include the drug group, study week, and drug group x study week interaction as predictors.

# 6. Exploratory Analysis

- a. We plan to examine the following biomarkers: MTHFR C677 CT/TT polymorphism, MTHFR A1298C polymorphism, FRa-autoantibody, and body mass index ≥30 kg/m²
  - i. Biomarkers are defined as typical or atypical based on standard values
  - ii. We will use mixed effects Poisson models to test the three-way interaction between drug group, study week, and biomarker. The outcome of interest will be the AISRS.